CLINICAL TRIAL: NCT04806945
Title: A Randomized, Double-blind, Placebo Controlled Phase III Study to Investigate Efficacy and Safety of First-Line Treatment With HLX10 (Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection) + Chemotherapy (Carboplatin/Cisplatin and Paclitaxel) vs Chemotherapy (Carboplatin/Cisplatin and Paclitaxel)in Patients With Advanced Cervical Cancer
Brief Title: A Phase III Study to Evaluate Efficacy and Safety of First-Line Treatment With HLX10 + Chemotherapy in Patients With Advanced Cervical Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor terminated the trial.
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-017-CC301
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX10 (Experimental): HLX10 + chemotherapy
  Interventions: Drug: HLX10; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin
- Placebo (Placebo Comparator): Placebo + chemotherapy
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Placebo to HLX10

INTERVENTIONS:
Drug: HLX10 — IV infusion.
  Other Names: Recombinant humanized anti-PD-1 monoclonal antibody injection
  Arms: HLX10
Drug: Paclitaxel — IV infusion
Drug: Cisplatin — IV infusion
Drug: Carboplatin — IV infusion
Drug: Placebo to HLX10 — IV infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of HLX10(Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection) plus chemotherapy compared to the efficacy and safety of placebo plus chemotherapy in the treatment of adult women with persistent, recurrent, or metastatic cervical cancer. Chemotherapy regimens include: paclitaxel plus cisplatin and paclitaxel plus carboplatin.

The primary study hypotheses are that the combination of HLX10 plus chemotherapy is superior to placebo plus chemotherapy with respect to: 1) Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as assessed by the IRRC or, 2) Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Has persistent, recurrent, or metastatic squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which has not been treated with systemic chemotherapy and is not amenable to curative treatment (such as with surgery and/or radiation)
2. CPS≥1
3. Has measurable disease per RECIST 1.1 as assessed by IRRC
4. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 14 days prior to randomization
5. Has adequate organ function

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
2. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years.
3. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
4. Has an active infection requiring systemic therapy
5. Has a known history of human immunodeficiency virus (HIV) infection
6. Has received prior therapy with an anti-PD-1, anti-PD-L1 or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4）

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cervical cancer only occurs in female.
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (assessed by the independent radiology review committee [IRRC] based on Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) | up to approximately 1 years
  Baseline until disease progression or death, whichever occurs first
Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: lingying wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No